CLINICAL TRIAL: NCT04056533
Title: Anti-CMV Pilot Clinical Trial: Prophylaxis of Cytomegalovirus Infection in Haploidentical Transplatation of Hematopoietic Progenitors With Adoptive Cell Inmunotherapy
Brief Title: Prophylaxis of Cytomegalovirus Infection With Adoptive Cell Inmunotherapy
Acronym: INMUNOCELL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INMUNOCELL
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: CMV
Keywords: Citomegalovirus; Haploidentical; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMV CTLs (Experimental): 1x10^5 CMV-CTLs/kg
  Interventions: Biological: CMV CTLs

INTERVENTIONS:
Biological: CMV CTLs — The donor derived cytomegalovirus specific T lymphocytes (CMV-CTL) will be transfused to the patients. The patients will receive CMV-CTL cells when their donors are sero-positive for CMV-DNA 21 days after transplant. The CMV-DNA levels will be monitored weekly for at least 100 days after the HAPLO. If after the initial dose of CMV-CTL cells the patient develops a viral infection, then they may be eligible to receive a CMV specific antiviral drug.

SUMMARY:
Cytomegalovirus (CMV) infection is a major cause of morbidity and mortality for recipients of allogeneic hematopoietic stem cell transplantation(HSCT). Recently, strategies based on immunotherapy adoptive cells (IAC) with anti-CMV Cytolitic T Lymphocytes (CMV-CTLs) has been incorporated to prevent or treat CMV after HSCT. The aim to study donor derived CMV-CTLs after haploidentical HSCT (HAPLO) as prophylaxis for CMV infection in transplant patients. CMV-CTLs will be administer at day 21 (+-7 days) post-HAPLO. CMV DNA levels with quantitative PCR will be weekly monitored.

DETAILED DESCRIPTION:
In HAPLO, CMV infection and disease are more frequent than in other type of HSCT, this is related to delayed immune reconstitution after transplant increasing post-transplant infectious complications. Approximately 60% of patients reactivated CMV infection after HAPLO and 15%, developed CMV disease afecting organs and causing the death of the patient in 8% of CMV disease cases.

If patient and donor are eligible, it will take 1x10^9 cells from donor leukapheresis. Donor cells will be selected and procesed by CliniMACs PRODIGY and after 12h it will obtain 7mL of CMV-CTLs. It will use 6mL of CMV-CTLs to infused a dose of 1x10^5 cells/kg in our patient. The donor derived CMV-CTL cells will be transfused into the patients' intravenous line. The patients will receive the dose of CMV-CTL cells when they are sero-positive for CMV-DNA 21 (+- 7 days) days after transplant.

The CMV-DNA levels will be monitored weekly for at least 100 days after the transplant. If after the initial dose of CMV-CTL cells the patient develops a viral infection, then the patient will receive treatment with anti-CMV comercial drugs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who received an alogeneic stem cell transplantation from haploidentical donors (HAPLO).
* Any source of stem cells (peripheral blood or bone marrow).
* CMV-seropositive donors.
* Negative pregnancy test in women.
* Signed writen informed consent.
* DONORS:

  1. HLA haploidentical and CMV-seropositve donors.
  2. Donor must be checked and suitable.
  3. Signed writen informed consent.
  4. Donor without active infection evidence at leukapheresis.

Exclusion Criteria:

* Patients without haploidentical CMV-seropositive donors.
* Patients who are not suitable for follow up visits.

CMV-CTLs Infusion Criteria:

* Hematopoiesis recovery at least partial (neutrophil counts >0.5x10^9/L in at least 3 consecutive samples post-transplant).

CMV-CTLs NON-Infusion Criteria:

* Patients receiving corticosteroid (dose of 0.5mg/kg/day of prednisone or equivalent) at infusion.
* ECOG > or = 3.
* Organic toxicities grade > or = 3.
* Patients who received ATG, donor lymphocytes or alemtuzuamb, 28 days pre-infusion.
* Patients with uncontroled infection defined by fevers and/or inestability and/or infection not resolved.
* Persistent fevers 3 days before infusion.
* Acute Graft Versus Host Disease (GVHD) grade II-IV.
* Relapse or progression after transplant and before infusion day.
* CMV reactivation/infection after transplant and before infusion day.

Patients who don´t fill infusion criteria, after day 28 post-HAPLO, will be considered screening failures and will be out of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
100-days incidence of CMV infection | From date of CMV-CTLs infusion to 100 days after transplant
  Viral load >200 copies in 1 sample

SECONDARY OUTCOMES:
1-year incidence of CMV specific antiviral drug use | From date of CMV-CTLs infusion to 1 year after transplant
  If viral load >200 copies in 2 samples or >1000 in 1 sample, treatment with valganciclovir will be started.
  Time from CMV-CTLs infusion until valganciclovir start and days of valganciclovir.
1-year incidence of CMV disease | From date of CMV-CTLs infusion to 1 year after transplant
  CMV disease P.Lungman criteria. CMV as primary cause of death.

OTHER OUTCOMES:
1-year incidence of CMV-CTLs adverse events | From date of CMV-CTLs infusion to 1 year after transplant
  Infusion reactions, causes of death, secondary graft failures and graft versus host disease (GVHD).
CMV-CTLs persistence | From date of CMV-CTLs infusion to 2 months after infusion
  Expansion of CMV-CTLs detected by flow cytometry.
Immune reconstitution post-HAPLO | From date of transplant to day 180 post-transplant
  CD3, CD4, CD8, B and NK lymphocyte counts in patient peripheral blood post-transplant (day 30, 60, 90 and 180) detected by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Galo Peralta Fernandez, MD, Study Director — Instituto de Investigación Marqués de Valdecilla
Locations (1):
- Hospital Marques de Valdecilla, Santander, Spain